CLINICAL TRIAL: NCT04945031
Title: The Study of Pharmacological Treatment Pattern for Cannabis-induced Psychosis
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: MU-DT/PY-IRB2019/PY114
Record Dates: First submitted 2021-06-15; First posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Cannabis
MeSH Terms: conditions — Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- cannabis-induced psychosis
  Interventions: Other: cannabis

INTERVENTIONS:
Other: cannabis — This study is observational study, we recorded history of substance used, symptoms and medication in a medical chart.

SUMMARY:
A cross-sectional and retrospective chart review study was conducted at the Princess Mother National Institute on Drug Abuse Treatment (PMNIDAT), Thailand. All patients who admitted at PMNIDAT from October 2013 to September 2019 were included. Patients aged 18-65 years who met the International Classification of Disease-10 (ICD-10) criteria of CIP and Had a positive urine test of cannabis were included. Cannabis use is a component cause of psychosis.More than half of symptoms of cannabis-induced psychosis (CIP) were hallucination, delusion, irritable and anxiety. Antipsychotic drug was still a key psychotropic drugs for treatment of CIP. However, antidepressants and benzodiazepines were commonly used for treatment of other symptoms beyond psychotics

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 12 years of age
* Patients who had been diagnosed as Cannabis-induced psychosis by International statistical Classification of Disease and Related Health problem (ICD-10) on 2016 code F12.5
* Patients had history of use of cannabis in medical chart
* Patients had the positive urine screening test of cannabis at the first day of admission

Exclusion Criteria:

* Patients had psychosis from organic psychosis, defined by diagnosis by ICD-10 code F09.6
* Unavailable data for evaluate of outcome especially data of drug use, content of drug use or urine screening test
* Patients who cancel of medical treatment before 7 day after admission.

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Medical chart which diagnosis by ICD-10 with cannabis-induced psychosis who admitted at PMNIDAT from October 2013 to September 2019 at Princess Mother National Institute on Drug Abuse Treatment.
Sampling Method: Non-Probability Sample
Enrollment: 317 (Actual)
Dates: Start 2019-11-08 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Pharmacological treatment pattern for cannabis-induced psychosis | 30 days
  Pharmacological treatment pattern for cannabis-induced psychosis during admission

SECONDARY OUTCOMES:
Change of Brief psychiatric rating scale (BPRS) form the first day of admission | Day1, Day 8, Day 15 and Day 22
  A high BPRS score is more severe of symptoms than a lower score

CONTACTS AND LOCATIONS:
Locations (1):
- Onrumpha Chuenchom, Thanyaburi, Changwat Pathum Thani, Thailand

REFERENCES:
- [Derived] Chuenchom O, Suansanae T, Lukanapichonchut L, Suwanmajo S, Suthisisang C. Real world clinical outcomes of treatment of cannabis-induced psychosis and prevalence of cannabis-related primary psychosis: a retrospective study. BMC Psychiatry. 2024 Sep 27;24(1):626. doi: 10.1186/s12888-024-06075-6. PMID 39334053